CLINICAL TRIAL: NCT00120055
Title: Association Between Systemic Exposure of Atorvastatin and Metabolites and Atorvastatin-induced Myotoxicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AVALIP04
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Myopathy
MeSH Terms: conditions — Muscular Diseases | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin (Lipitor)

SUMMARY:
The aim of this study is to investigate whether the pharmacokinetics of atorvastatin and/or its metabolites is altered in patients with confirmed atorvastatin-induced myopathy compared to healthy controls.

DETAILED DESCRIPTION:
A 24 hour pharmacokinetic investigation of atorvastatin and metabolites will be performed in 15 patients with a history of atorvastatin -induced myotoxicity. The possible link to relevant mutations in SLCO1B1, CYP3A5 and MDR1 will be also be investigated

ELIGIBILITY:
Inclusion Criteria:

* above 18 years
* previous history of atorvastatin-associated myotoxicity

Exclusion Criteria:

* current treatment with drugs or herbal remedies with known pharmacokinetic interaction potential with atorvastatin
* previous CK levels above ten times the upper limit of normal range
* pregnancy and persistent muscular complaints after a four week wash-out period of statin treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2005-04

PRIMARY OUTCOMES:
Statin toxicity | 1 year
  Rechallenge test of statin induce toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, PhD, Study Chair — University of Oslo School of Pharmacy